CLINICAL TRIAL: NCT05797337
Title: Knowledge and Attitude of Dialysis Center Medical Staff Towards Living Kidney Donation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Paulina Kurleto, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: WLNZ/NoZ/3/2023
Record Dates: First submitted 2023-02-28; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cross-sectional study is to learn about the level of knowledge and attitudes of medical staff working in dialysis centers about living kidney donations. The main questions it aims to answer are:

* What is the level of knowledge of dialysis center medical staff regarding living kidney transplantations?
* How much time does the staff have for educating the patients about living kidney donations? Participants will be asked to answer a self-report questionnaire along with two standardized tools.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent to participate in the study.
* Communicative knowledge of the Polish language.
* Each potential participant will receive comprehensive information about the purpose and course of the study before participating in the study and will consent to the study.
* Dialysis station employee: doctor, nurse.

Exclusion Criteria:

* no consent
* no communicative knowledge of the Polish language
* not working in dialysis center currently

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dialysis center workers (doctors, nurses)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge and attitudes of dialysis centers medical workers toward living kidney donations. | 22 months
  Knowledge and attitudes will be measured using a 38-item self-report questionnaire with single and multi-choice questions.
How satisfaction with life impacts attitudes toward living kidney donation | 22 months
  Polish adaptations of a standardized tool will be used to measure satisfaction with life.
  Satisfaction with Life Scale with responses measured using a 7-point Likert scale, where: 7-I strongly agree, 6-I agree, 5-I tend to agree, 4-I neither agree nor disagree, 3-I tend to disagree, 2-I disagree, 1-I strongly disagree. The result of the measurement was a general indicator of the feeling of satisfaction with life ranging from 5 to 35 points (scores of 20 are considered neutral).
How self-esteem impacts attitudes toward living kidney donation | 22 months
  Polish adaptations of standardized tools will be used to measure self-esteem.
  A 10-item Rosenberg Self-Esteem Scale (RSES) with responses measured on a 4-item Likert scale where: 0 (strongly agree), 1 (agree), 2 (disagree), and 3 (strongly disagree). The maximum score is 30, and higher scores indicate higher self-esteem.
How empathy impacts attitudes toward living kidney donation | 22 months
  Polish adaptations of standardized tools will be used to measure empathy.
  Davis' Interpersonal Reactivity Index (IRI), a 28-item self-report questionnaire using a 5-item Likert scale with two anchors (A=Does not describe me well; E=Describes me very well). The IRI covers multiple dimensions of empathy.
How self-efficacy impacts attitudes toward living kidney donation | 22 monts
  Polish adaptations of standardized tools will be used to measure self-efficacy.
  General Self-Efficacy Scale (GSE) with the total score calculated by finding the sum of all the items and ranges between 10 and 40, with a higher score indicating more self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrzej Frycz Modrzewski Krakow University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided